CLINICAL TRIAL: NCT04254172
Title: A SINGLE-SITE, PROSPECTIVE, NATURAL HISTORY LOW INTERVENTIONAL STUDY TO ESTABLISH NORMATIVE DATA OF REAL-WORLD ACTIVITY MEASURES USING WEARABLE SENSORS IN AMBULATORY BOYS WITH DUCHENNE MUSCULAR DYSTROPHY (DMD)
Brief Title: A Low Interventional Study to Monitor Activity Using Wearable Sensors in Duchenne Muscular Dystrophy
Status: Terminated | Type: Observational
Why Stopped: This low-interventional study (involving no study drug) has been terminated early due to the COVID-19 pandemic, and not for any safety or efficacy reasons.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3391005
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Fitness Trackers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Single cohort: There is no randomization or stratification in this study. All subjects will complete the same study assessments.
  Interventions: Device: Activity Monitor

INTERVENTIONS:
Device: Activity Monitor — Wrist and ankle sensors to be worn continuously for 2-week intervals.

SUMMARY:
The purpose of this low interventional study is to collect data on everyday movement in boys with Duchenne muscular dystrophy (DMD) using wearable activity sensors. The activity sensors could provide useful information beyond what is currently collected by functional (movement, strength) assessments in clinic. This information can help with the understanding of the impact of DMD, and perhaps with how possible treatments can affect this impact.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Duchenne muscular dystrophy confirmed by medical history and genetic testing
* Body weight between 15 and 50 kg
* Receipt of glucocorticoids for 6 months and a stable daily dose for at least 3 months prior to study entry
* Ability to rise from floor within seven (7) seconds and ability to walk

Exclusion Criteria:

* Current exposure to systemic immunosuppressant agents other than glucocorticoids.
* Prior exposure to any gene therapy agent, including exon-skipping and missense agents.
* Exposure to other investigational drugs within 30 days or 5 half-lives, whichever is longer.
* Any injury which may impact functional testing per investigator's judgement. Previous injuries must be fully healed prior to consenting. Prior lower limb fractures must be fully healed and at least 3 months from injury date at screening.
* Any planned surgeries which may impact physical activity and performance.
* Presence or history of musculoskeletal or neurological disease in addition to DMD.
* Any known allergies or skin reactions to stainless steel, versaflex, and silicon that may cause possible discomfort by wearable sensors.
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, cancer, autoimmune or allergic disease that may interfere with the study conduct as per investigator's judgment, excluding untreated, asymptomatic, seasonal allergies at time of screening.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are Pfizer employees, including their family members, directly involved in the conduct of the study.

Ages: 4 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Study Population: Ambulatory boys with Duchenne muscular dystrophy who receive care at Nationwide Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline and variability of activity measures | baseline, 3, 6, 9, and 12 months

SECONDARY OUTCOMES:
Mean change from baseline in functional assessment scores obtained in the clinic | baseline, 3, 6, 9, and 12 months
Comparison of mean changes from baseline and correlation coefficient between activity monitoring data and functional data obtained in clinic | baseline, 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3391005